CLINICAL TRIAL: NCT01374633
Title: Effect on Sevoflurane Sedation on Intra Cranial Pressure in Traumatic Brain Injury Patients
Brief Title: Sevoflurane Sedation on Intra Cranial Pressure in Traumatic Brain Injury Patients
Acronym: SEPIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100206; 2011-000253-23 (Other: Eudra CT)
Record Dates: First submitted 2011-06-08; First posted 2011-06-16 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Brain Injury
Keywords: Sevoflurane; Brain injury; Intra cranial pressure; Sedation; Brain injury with initial Glasgow score less than 9
MeSH Terms: conditions — Brain Injuries | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1:patient with severe traumatic brain (Experimental)
  Interventions: Drug: 1: Sevoflurane

INTERVENTIONS:
Drug: 1: Sevoflurane — Mean sevoflurane infusion rate will be around 6 ml/h or 72 ml for 12 hours. Maximal infusion rate will be around 12 ml/h, or 144 ml for 12 hours. Packaging: bottle containing 250 ml of liquid sevoflurane for evaporation. Administration mode: anaesthetic conserving device for volatile anaesthetics."
  Other Names: SEVORANE (Abbott); SEVOFLURANE (Baxter)

SUMMARY:
Main purpose of the study is to evaluate the effect of sevoflurane on intra cranial pressure (ICP) after traumatic brain injury. Patients admitted for traumatic brain injury equipped with ICP measurement will be sedated with sevoflurane via the Anaconda device during 12 hours. Sedation will be controlled with BIS.

DETAILED DESCRIPTION:
Sedation is most of the time required for ICP management after traumatic brain injury. Sevoflurane, an inhaled anaesthetic drug is commonly used in operatory room. Thanks to a new device, the Anaconda, it now can be applied to intensive care patients. His advantages a rapid elimination after administration stops, which can allow an early neurologic evaluation, very important for traumatic brain injury patients.We will study the effect of sevoflurane administration on ICP of TBI patients. Patients admitted for severe TBI (Glasgow come scale < 8), equipped with ICP sensor, elder than 18 years old will be include. A sedation with sevoflurane will be administrated during 12 hours instead of classical intra venous sedation with midazolam, depending on BIS score. ICP evolution will be characterised in success if < 30 mmHg or failure if ≥ 30 mmHg.6 patients will be included for the first phase. The study will be stopped if the failures are ≥ 2. Otherwise, 27 patients will be included. Study will be stopped if failures number ≥ 5 before the end if the inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* severe traumatic brain injury (glasgow < 8)
* age > 18
* no surgery scheduled
* sedation with midazolam and sufentanil
* ICP sensor

Exclusion Criteria:

* external ventricular derivation
* pregnancy
* antecedent of malign hyperthermia
* haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
ICP evolution | ICP will be continuously recorded during the 12 hours of sedation with sevoflurane
  patients where ICP increase more than 30 mmHg during more than 15 minutes will be characterized as "failure". Patients whose ICP do not increase during the 12 hours of sedation with sevoflurane will be characterized as "success".

SECONDARY OUTCOMES:
Sedation level | during the 12 hours of sedation with sevoflurane
  sedation level will be evaluated with the measure of the Bispectral Index and the SAS sedation score. Proportion of time with BIS of 45-65% and SAS <2, which are the objective of sedation level, will be recorded.
Haemodynamic tolerance | during the 12 hours of sedation with sevoflurane
  invasive mean arterial pressure (MAP) will be continuously recorded. Hypotension is defined by a MAP less than 60 mmHg.
Malignant hyperthermia screening | during the 12 hours of sedation with sevoflurane
  increase of eardrum temperature more than 39°C is considered as potential malignant hyperthermia

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DURANTEAU, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Reanimation Chirurgicale - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre, France